CLINICAL TRIAL: NCT01460134
Title: A Phase 1, Open-label, Dose-escalation, Safety and Pharmacokinetic Study of CDX-1127 in Patients With Selected Refractory or Relapsed Hematologic Malignancies or Solid Tumors
Brief Title: A Study of CDX-1127 (Varlilumab) in Patients With Select Solid Tumor Types or Hematologic Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDX1127-01
Record Dates: First submitted 2011-10-12; First posted 2011-10-26 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2017-08

CONDITIONS: CD27 Expressing B-cell Malignancies for Example Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia; Mantle Cell Lymphoma; Marginal Zone B Cell Lymphoma); Any T-cell Malignancy; Solid Tumors (Metastatic Melanoma, Renal (Clear) Cell Carcinoma; Hormone-refractory Prostate Adenocarcinoma, Ovarian Cancer; Colorectal Adenocarcinoma, Non-small Cell Lung Cancer); Burkett's Lymphoma; Primary Lymphoma of the Central Nervous System
Keywords: CD27 expressing Hematologic Malignancies; CD27 expressing Solid Tumors; chronic lymphocytic leukemia; Burkett's lymphoma; mantle cell lymphoma; primary lymphoma of the central nervous system; marginal zone B cell lymphoma; solid tumor; metastatic melanoma; renal (clear) cell carcinoma; hormone-refractory prostate adenocarcinoma; ovarian cancer; colorectal adenocarcinoma; non-small cell lung cancer
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Melanoma; Margins of Excision; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell | interventions — varlilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Hematologic Malignancies (Dose Escalation) (Experimental): B-Cell Enrollment COMPLETED T-Cell Enrollment COMPLETED
  Interventions: Drug: CDX-1127
- Solid tumors (Dose Escalation; COMPLETED) (Experimental)
  Interventions: Drug: CDX-1127
- Solid Tumors (Expansion Phase; COMPLETED) (Experimental): Several expansion cohorts of up to 15 patients each are planned, including melanoma and renal cell carcinoma.
  Interventions: Drug: CDX-1127
- Hematologic Malignancies (COMPLETED) (Experimental): Several expansion cohorts of up to 15 patients each are planned, including Hodgkin lymphoma.
  Interventions: Drug: CDX-1127

INTERVENTIONS:
Drug: CDX-1127 — Patients will initially receive a single dose of CDX-1127, followed by a 28-day observation period and a Multi-Dose Phase (one "cycle" of 4 weekly doses of CDX-1127). All patients with stable disease who do not experience a DLT or start alternate anti-cancer treatments may then be eligible for a Retreatment Phase (up to 4 additional "cycles"). Patients with confirmed partial response or complete response will be followed for response duration and may be eligible for additional cycles of treatment at the time of relapse/progression.
  The dose of CDX-1127 given for the Dose Escalation phase will depend on the cohort each patient is assigned to, and will range between 0.1 and 10.0 mg/kg of CDX-1127.
  Arms: Hematologic Malignancies (Dose Escalation); Solid tumors (Dose Escalation; COMPLETED)
Drug: CDX-1127 — Patients will receive 4 weekly doses of CDX-1127 followed by an observation period. All patients with stable disease who do not experience a DLT or start alternate anti-cancer treatments may then be eligible for a Retreatment Phase (up to 4 additional "cycles"). Patients with confirmed partial response or complete response will be followed for response duration and may be eligible for additional cycles of treatment at the time of relapse/progression.
  Arms: Solid Tumors (Expansion Phase; COMPLETED)
Drug: CDX-1127 — Patients will receive four doses of CDX-1127 administered every three weeks followed by an observation period. All patients with stable disease who do not experience a DLT or start alternate anti-cancer treatments may then be eligible for a Retreatment Phase (up to 4 additional "cycles"). Patients with confirmed partial response or complete response will be followed for response duration and may be eligible for additional cycles of treatment at the time of relapse/progression.
  Arms: Hematologic Malignancies (COMPLETED)

SUMMARY:
This is a study of CDX-1127, a therapy that targets the immune system and may act to promote anti-cancer effects. The study enrolls patients with hematologic cancers (certain leukemias and lymphomas), as well as patients with select types of solid tumors.

DETAILED DESCRIPTION:
CDX-1127 is a fully human monoclonal antibody that binds to a molecule called CD27 found on certain immune cells and also on certain hematologic tumor cells and may act to promote anti-tumor effects.

This study will evaluate the safety and activity of escalating doses of CDX-1127 in patients with B-cell and T-cell hematologic malignancies known to express CD27 and solid tumors that are more likely to be responsive to the immune system.

Eligible patients who enroll in the dose escalation portion of the study will be assigned to one of 5 dose levels of CDX-1127. This first phase of the study will test the safety profile of CDX-1127 and will assess which dose to test in future studies.

During the Expansion phase, cohorts of approximately 15 patients each will receive the study treatment to continue to evaluate the safety profile of CDX-1127 and to determine if it has an effect on their cancer. Expansion cohorts may be limited to one or more tumor types.

Patients enrolled in the study may receive study treatment for up to 5 cycles, until their disease has progressed or until it is necessary to stop the treatment for safety or other reasons.

All patients enrolled in the study will be closely monitored to determine if their cancer is responding to treatment and for any side effects that may occur.

ELIGIBILITY:
Inclusion Criteria:

Among other criteria, patients must meet the following conditions to be eligible for the study:

1. 18 years of age or older.
2. Body Weight ≤ 120 kg.
3. Histologic diagnosis of either a B-cell or T-cell hematologic malignancy known to express CD27 or one of the following solid tumors: metastatic melanoma, renal (clear) cell carcinoma, hormone-refractory prostate adenocarcinoma, ovarian cancer, colorectal adenocarcinoma or non-small cell lung cancer. For the solid tumor expansion cohorts, enrollment is limited to the following solid tumors: melanoma and renal cell carcinoma.
4. Tumor must be recurrent or treatment refractory with no remaining alternative, approved therapy options, with the following exception: melanoma patients enrolled in the expansion phase must have previously received ipilimumab and, for patients with the BRAF V600E mutation, vemurafenib, or have been offered such therapies and refused, and patients must have progressive disease subsequent to previous therapies.
5. Measurable or evaluable disease.
6. Have adequate blood, bone marrow, liver and kidney function as determined by laboratory tests.
7. If of childbearing potential (male or female), agree to practice an effective form of contraception during study treatment.
8. Have little or no side effects remaining from prior cancer therapies.
9. Provide written informed consent.

Exclusion Criteria:

Among other criteria, patients who meet the following conditions are NOT eligible for the study:

1. Known prior primary or metastatic brain or meningeal tumors.
2. Receiving treatment with immunosuppressive agents, including any systemic steroids.
3. Active infection requiring systemic therapy, known HIV infection, or positive test for hepatitis B surface antigen or hepatitis C.
4. Is being treated for anti-coagulation (i.e. warfarin) for reasons other than catheter patency.
5. Women who are pregnant or lactating.
6. Prior allogeneic bone marrow transplant.
7. Autologous bone marrow transplant within 100 days of first dosing.
8. Recent chemotherapy or other anti-cancer therapy (within 2 - 14 weeks depending on treatment type).
9. Systemic radiation therapy within 4 weeks or prior focal radiotherapy within 2 weeks prior to first dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-10; Primary Completion 2015-12 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Characterize the adverse events associated with CDX-1127 administration | Safety follow up is 70 days from last dose.
  Analysis of adverse events along with the results of vital sign measurements, physical examinations, and clinical laboratory tests will be used to determine the safety profile of CDX-1127.

SECONDARY OUTCOMES:
Levels of anti-CD27 antibodies in circulating blood. | Until end of treatment
Levels of CDX-1127 in circulating blood. | Until end of treatment
Activity Evaluations | Until disease progression
  Determine the anti-malignant cell activity of CDX-1127 based on change from baseline in tumor measurements every 12 weeks.
Immune system effects (eg: lymphoid cell populations and serum cytokine levels) | Until end of treatment

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Mayo Clinic Arizona - Cancer Clinical Research Unit, Scottsdale, Arizona
  - Stanford Cancer Center - Stanford University, Stanford, California
  - Mayo Clinic, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai Hess Center for Science and Medicine, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research Centers - Medical City, Dallas, Texas
  - University of Virginia Health System, Charlottesville, Virginia

REFERENCES:
- [Background] Burris HA, Infante JR, Ansell SM, Nemunaitis JJ, Weiss GR, Villalobos VM, Sikic BI, Taylor MH, Northfelt DW, Carson WE 3rd, Hawthorne TR, Davis TA, Yellin MJ, Keler T, Bullock T. Safety and Activity of Varlilumab, a Novel and First-in-Class Agonist Anti-CD27 Antibody, in Patients With Advanced Solid Tumors. J Clin Oncol. 2017 Jun 20;35(18):2028-2036. doi: 10.1200/JCO.2016.70.1508. Epub 2017 May 2. PMID 28463630
- [Derived] Ansell SM, Flinn I, Taylor MH, Sikic BI, Brody J, Nemunaitis J, Feldman A, Hawthorne TR, Rawls T, Keler T, Yellin MJ. Safety and activity of varlilumab, a novel and first-in-class agonist anti-CD27 antibody, for hematologic malignancies. Blood Adv. 2020 May 12;4(9):1917-1926. doi: 10.1182/bloodadvances.2019001079. PMID 32380537